CLINICAL TRIAL: NCT04148079
Title: Frequency of Arrhythmias During Physiotherapy
Brief Title: Safety of Electrotherapy in Patients With Knee Osteoarthritis and Cardiac Diseases
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ciubean Alina Deniza, Principal investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: UniversitateaMFH
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical therapy — low frequency currents (galvanic or TENS), medium frequency currents (interferential) and high frequency currents (short wave diathermy), all combined with an individualized exercise program and massage therapy

SUMMARY:
This study aimed to asses whether physyical therapy (e.g. electrotherapy in the form of low, medium or high frequency currents, massage and kinetotherapy) for treatment of knee osteoarthritis can induce or aggravate certain cardiac diseases during or immediately after therapy. The physyical treatment described is not a new method, is currently used and recommended in all guidelines for non-pharmacological and non-surgical therapy of knee osteoarthritis. What is not clear is whether application of electrotherapy in the knee area can alter the preexisting cardiac condition.

DETAILED DESCRIPTION:
An analytical and transversal study was carried out between March 2013 and August 2017. The study included a total of 46 patients previously diagnosed with degenerative knee OA. All the patients included in the study were recruited during inpatient visit in the Clinical Rehabilitation Hospital in Cluj-Napoca, Romania.

Each patient was clinically evaluated and was furthermore prescribed a PT program (ET, massage and kinesiotherapy). They were monitored by 24 hour-Holter ECG in 2 separate days, at the beginning of treatment, before applying the PT methods (day 1), and after completing a 10-day PT program (day 2).

PT modalities prescribed for each patient after clinical evaluation included different types of ET, all currently used and included in the national and international treatment guidelines, as in low frequency currents (galvanic or TENS), medium frequency currents (interferential) and high frequency currents (short wave diathermy), all combined with an individualized exercise program and massage therapy. The program was performed on a daily basis, for 10 days.

The aim of the PT program was to decrease pain and increase range of motion in the affected joints and did not lead to increases in cardiac frequencies. No hydrotherapy was applied, given that that the Holter ECG was not waterproof. No technical incidents were reported during the study. No alternate positioning of the patient wearing a Holter ECG for ET procedures was necessary, as the region of interest was the knee. No change in current drug therapy was allowed for the whole duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis and imaging diagnosis of knee osteoarthrtitis based on ACR 2000 diagnostic criteria

Exclusion Criteria:

* known cardiac arrhythmias (atrial fibrillation, atrial flutter)
* congestive heart failure class NYHA II, III or IV
* any other general contraindications for PT (infections, psychiatric disorders etc)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 46 patients, 33 female, 13 male 20 patients had a history of arrythmias (e.g.premature atrial contractions) 19 patients had a history of ischemic heart disease
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from Baseline after 10 days
  Minimal, average, maximum heart rate evaluated by 24 hour Holter EKG monitoring
Supraventricular, ventricular and total Extrasystoles | Change from Baseline after 10 days
  supraventricular, ventricular, total extraystoles evaluated by 24 hour Holter EKG monitoring

IPD SHARING:
Plan to Share IPD: Undecided
If asked for the data from someone who needs it, we will be happy to share